CLINICAL TRIAL: NCT03838354
Title: A Prospective, Multicenter Clinical Trial of Chidamide in the Management of Refractory Immune Thrombocytopenia
Brief Title: A Clinical Trial of Chidamide in the Management of Refractory ITP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Chidamide
Record Dates: First submitted 2018-11-27; First posted 2019-02-12 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Thrombocytopenia
Keywords: ITP; Chidamide
MeSH Terms: conditions — Thrombocytopenia | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; HBI-8000

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Chidamide 2.5 mg po twice per week
  Interventions: Drug: Chidamide
- B (Experimental): Chidamide 5 mg po twice per week
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — In the 2.5 mg group, chidamide will be administered orally at an initial dose of 2.5 mg twice per week for 12 weeks. If an initial response was achieved by week 12, the allocated treatment could continue. Patients in 2.5 mg group were allowed to increase dose to 5 mg if platelet counts were less than 30×10^9 cells per L or less than two-times increase from baseline platelet count at week 12 according to investigators' advice and the patients' decision.
  Other Names: HBI-8000
  Arms: A
Drug: Chidamide — In the 5 mg group, chidamide will be administered orally at an initial dose of 5 mg twice per week for 12 weeks. If an initial response was achieved by week 12, the allocated treatment could continue. Patients who did not respond to chidamide at 5 mg for 12 weeks would stop the allocated treatment and were continuously followed up.
  Other Names: HBI-8000
  Arms: B

SUMMARY:
Primary immune thrombocytopenia (ITP) is an autoimmune bleeding disorder. Increased macrophage phagocytosis of antibody-coated platelet as well as decreased number and/or impaired function of CD4+CD25+Foxp3+ regulatory T (Treg) cells have been shown to participate in the pathogenesis of ITP. Our preclinical data revealed that chidamide, a histone deacetylase inhibitor (HDACi), could attenuate macrophage phagocytosis of antibody-coated platelets, stimulate production of natural Foxp3+ Tregs, and upregulate CTLA4 expression through modulation of histone H3K27 acetylation. The project was undertaking by Qilu Hospital of Shandong University in China. In order to evaluate the efficacy and safety of chidamide at two different dosage regimens in adult patients with refractory ITP.

DETAILED DESCRIPTION:
In this prospective, open-label, multicenter, randomized clinical trial, refractory ITP adult patients will be enrolled from five medical centers in China. Eligible participants will be randomly assigned 1:1 to receive chidamide at either 2.5 or 5 mg twice per week. The primary endpoint is the overall response at week 12. Complete response was defined as a platelet count at or above 100×10^9/L and an absence of bleeding. Partial response was defined as a platelet count at or above 30×10^9/L but less than 100×10^9/L and at least a doubling of the baseline platelet count and an absence of bleeding. No response was defined as a platelet count of less than 30×10^9 cells per L, or less than two-times increase from baseline platelet count, or bleeding. The secondary enpoints included 6-month sustained response, time to response (TTR), duration of response, bleeding scores, health-related quality of life assessment and adverse events (AEs). This study will compare the efficacy and safety of chidamide in two different dosage regimens in adult patients with refractory.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of the screening.
* Participant may be male or female.
* Participant has a confirmed diagnosis of ITP according to the 2019 International Working Group assessment for more than 6 months at screening.
* Participant who didn't respond or relapsed after previous first-line treatment, and lack of response to rituximab, TPO agents, or splenectomy.
* Bone marrow biopsy is performed in participants over 60 years to exclude hematological malignancies.

Exclusion Criteria:

* Participant has evidence of a secondary cause of immune thrombocytopenia or to drug treatments or participant has a multiple immune cytopenia, e.g. Evan's syndrome.
* Participant with the following conditions:severe dysfunction of the heart, kidney, liver, or lung; severe immunodeficiency; malignancy; HIV; hepatitis B or C virus infection; pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Overall response at week 12 | week 12
  The primary endpoint was the overall response at week 12.Complete response was defined as a platelet count at or above 100×10^9/L and an absence of bleeding. Partial response was defined as a platelet count at or above 30×109/L but less than 100×10^9/L and at least a doubling of the baseline platelet count and an absence of bleeding. No response was defined as a platelet count of less than 30×10^9 cells per L, or less than two-times increase from baseline platelet count, or bleeding.

SECONDARY OUTCOMES:
Therapy associated adverse events | up to 1 year per subject
  The number and frequency of therapy associated adverse events
Sustained response | 6 months
  A response lasting for at least 6 months was defined as a sustained response.
Time to response | 12 weeks
  Time to response was defined as the time from treatment initiation to achieve a complete response or a partial response, whichever came first, assessed up to week 12.
Duration of response | 12 months
  Duration of response was defined as the time from achievement of a complete response or a partial response to the loss of response.
Bleeding scores | 12 months
  Bleeding symptoms were graded according a standardized bleeding scale specific to primary immune thrombocytopenia on the basis of site and severity of bleeding by Khellaf et al (PMID: 15951296). A modification was made to exclude age from the original scale so that only bleeding symptoms were described. At each visit, we recorded bleeding scores. Routine visits were scheduled once a week for the first 4 weeks and once a month thereafter. Scores ranged from 0 to 59, with higher values indicating higher bleeding risk.
Health-related quality of life assessment | 12 weeks
  Health-related quality of life was assessed using a self-administered immune thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) at baseline and at week 12. Scores ranged from 0 to 100, with higher values indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China